CLINICAL TRIAL: NCT04191044
Title: Portal Hypertension in Non-alcoholic Fatty Liver Disease: Association With Cardiovascular Risk and Identification of Non-invasive Biomarkers
Brief Title: Portal Hypertension in Non-alcoholic Fatty Liver Disease: Association With Cardiovascular Risk and Identification of Non-invasive Biomarkers (THESIS)
Acronym: THESIS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Collaborators: Hospital Universitario Ramon y Cajal (Other); Hospital General Universitario Gregorio Marañon (Other); Puerta de Hierro University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: THESIS
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Fatty Liver Disease
Keywords: Non-alcoholic fatty liver disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be used to measure inflammation markers and other laboratory parameters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- NAFLD with mild steatosis and grade <3 fibrosis in patients: NAFLD with mild steatosis and grade <3 fibrosis in patients with grade 1 or 2 obesity and insulin resistance (HOMA index> 2.6) or diabetes mellitus.
  Interventions: Other: A complete cardiovascular and liver characterization will be carried out
- NAFLD with severe steatosis and grade <3 fibrosis in patients: NAFLD with severe steatosis and grade <3 fibrosis in patients with grade 1 or 2 obesity and insulin resistance (HOMA index> 2.6) or diabetes mellitus.
  Interventions: Other: A complete cardiovascular and liver characterization will be carried out
- NAFLD with advanced fibrosis: NAFLD with advanced fibrosis (i.e. grade 3 or 4 fibrosis) without previous portal hypertension-related complications
  Interventions: Other: A complete cardiovascular and liver characterization will be carried out
- Decompensated NAFLD cirrhosis: Decompensated NAFLD cirrhosis (i.e. development of ascites, variceal hemorrhage, and/or hepatic encephalopathy) up to Child B (9 points)
  Interventions: Other: A complete cardiovascular and liver characterization will be carried out

INTERVENTIONS:
Other: A complete cardiovascular and liver characterization will be carried out — A complete cardiovascular and liver characterization will be carried out, including some supplementary tests with minimal risks (e.g. hemodynamic study). If any disease is detected, patients will be referred to the corresponding specialized care following the usual clinical practice.

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is the most frequent cause of chronic liver disease in our environment. Preliminary data suggest that portal hypertension may exist in the initial phases of NAFLD due to mechanisms that have not yet been elucidated. The clinical relevance of its development in these initial phases is unknown, while in more advanced phases new data are required to confirm the close relationship between portal hypertension and the risk of decompensation described in other etiologies. Likewise, the influence of fibrosis and portal hypertension on the cardiovascular risk of patients with NAFLD is unknown. The aim of the present multicenter project is to characterize the presence of portal hypertension and the mechanisms involved in its development in the different stages of NAFLD, to assess the association between the degree of portal hypertension and the development of portal hypertension-related complications, to know the early cardiovascular risk in the different stages of the disease, and to identify noninvasive biomarkers of the presence and severity of portal hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Clinical suspicion of NAFLD.
* Severe (controlled attenuation parameter (CAP) ≥330 dB/m) or mild steatosis (CAP: 298-317 dB / m), and FibroScan® grade 2 fibrosis (M probe: 7-9 kpa; XL probe: 5-7.5 kpa) in patients with grade 1 or 2 obesity and insulin resistance (HOMA index> 2.6) or diabetes mellitus.
* Fibroscan® grade 3 or 4 fibrosis (M probe:> 9 kpa; XL probe:> 7.5 kpa).
* Decompensated NAFLD cirrhosis (i.e. development of ascites, variceal hemorrhage, and/or hepatic encephalopathy) up to Child B (9 points).
* Signature of informed consent.

Exclusion Criteria:

* Concomitant liver disease and patients with acute on chronic liver failure.
* Excessive alcohol consumption (≥ 30 grams per day in men and ≥ 20 grams per day in women).
* Comorbidities (HIV infection, connective diseases, prothrombotic disorders) and/or drugs (didanosine, azathioprine, oxaliplatin) associated with the presence of idiopathic non-cirrhotic portal hypertension.
* Clinical history of cardiovascular disease (ischemic cardiomyopathy, atrial fibrillation, valvular defects, severe arterial hypertension, previous hospitalizations secondary to heart failure, cerebrovascular disease).
* Severe renal impairment, defined by creatinine clearance <15 ml/min/1.73m2.
* Any previous or current thrombosis in any venous territory.
* Uncontrolled psychiatric illness
* Contraindication to liver biopsy or any of the complementary tests included in the project.
* Hepatocellular carcinoma that does not meet Milan criteria.
* Pregnancy or breastfeeding
* Significant comorbidities that entail a functional limitation and/or a life expectancy of less than 12 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-alcoholic fatty liver disease.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2020-01-10 (Estimated); Primary Completion 2020-01-10 (Estimated); Study Completion 2020-07-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with NAFLD without advanced fibrosis and severe steatosis with portal hypertension | 1 months
Number of patients with NAFLD and advanced fibrosis with portal hypertension | 1 months
number of the mechanisms responsible for the appearance of portal hypertension by specifically assessing the following | 1 months
  An increase in sinusoidal vascular resistance and the relative importance of its structural (sinusoidal compression) and functional (endothelial dysfunction and activation of starry cells) components, Splanchnic vasodilatation leading to portal hyperflow and hyperdynamic circulation, proinflammatory state and Activation of angiogenesis.
Threshold of portal hypertension leading to portal hypertension-related complications in patients with NAFLD | 1months

SECONDARY OUTCOMES:
Impact of portal hypertension and hepatic fibrosis on early cardiovascular risk and the degree of liver and kidney function. | 1 months
Non-invasive biomarkers of the presence and severity of portal hypertension through metabolomics, extracellular vesicles and / or other analytical markers | 1 months
  liquid biopsy

REFERENCES:
- [Background] Baffy G. Origins of Portal Hypertension in Nonalcoholic Fatty Liver Disease. Dig Dis Sci. 2018 Mar;63(3):563-576. doi: 10.1007/s10620-017-4903-5. Epub 2018 Jan 22. PMID 29368124
- [Background] Francque S, Verrijken A, Mertens I, Hubens G, Van Marck E, Pelckmans P, Van Gaal L, Michielsen P. Noncirrhotic human nonalcoholic fatty liver disease induces portal hypertension in relation to the histological degree of steatosis. Eur J Gastroenterol Hepatol. 2010 Dec;22(12):1449-57. doi: 10.1097/MEG.0b013e32833f14a1. PMID 21389796
- [Background] Mendes FD, Suzuki A, Sanderson SO, Lindor KD, Angulo P. Prevalence and indicators of portal hypertension in patients with nonalcoholic fatty liver disease. Clin Gastroenterol Hepatol. 2012 Sep;10(9):1028-33.e2. doi: 10.1016/j.cgh.2012.05.008. Epub 2012 May 18. PMID 22610002
- [Background] Rodrigues SG, Montani M, Guixe-Muntet S, De Gottardi A, Berzigotti A, Bosch J. Patients With Signs of Advanced Liver Disease and Clinically Significant Portal Hypertension Do Not Necessarily Have Cirrhosis. Clin Gastroenterol Hepatol. 2019 Sep;17(10):2101-2109.e1. doi: 10.1016/j.cgh.2018.12.038. Epub 2019 Jan 6. PMID 30625404